CLINICAL TRIAL: NCT06127277
Title: Next4You: : A Fully Mobile Relationships Based Program for Youth in Foster Care
Brief Title: Next4You: A Fully Mobile Relationships Based Program for Youth in Foster Care
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: ETR Associates (Other)
Collaborators: RTI International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Next4You
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Pregnancy Related; Adolescent Behavior; Sexually Transmitted Diseases
Keywords: Pregnancy; Adolescence; Sexually Transmitted Infections; Decision Making; Prevention Education
MeSH Terms: conditions — Adolescent Behavior; Sexually Transmitted Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Next4You (Experimental): Next4You is a web-based, self-paced program featuring 6 content modules, each containing 8-10 microlessons intended to reduce rates of unintended pregnancy and sexually transmitted infections (STI) and increase essential knowledge, attitudes, and skills among young people aged 16-19 currently in foster care in California. Each microlesson is 2-4 minutes with diverse content formats. Youth in the intervention condition will have unlimited access to the platform for an intensive 4-week period. During this period, engagement activities will be deployed twice weekly to draw users back into the platform for further engagement with the microlessons. Content will also be released on a schedule to encourage continued engagement. Following the intensive 4-week period, youth will retain unlimited access to the platform but will not receive reminders to engage with the content. Participants complete online surveys at baseline, as well as 3 months and 9 months after the intervention ends.
  Interventions: Behavioral: Next4You
- General Health Mobile Website (Active Comparator): Youth randomized to the attention control condition will have access to a mobile-responsive website that contains digital resources focusing on nutrition, sleep, stress/anxiety, and exercise. Like the intervention group, participants in the attention control group will have unlimited access to the general health digital resources for an intensive 4-week period. Each topic area will have between 1-4 digital pamphlets (for a total of 12 pamphlets) that are downloadable and take between 2-4 minutes to read. Participants complete online surveys related to attitudes, knowledge, and behavior around romantic relationships and sexual behavior at baseline, as well as 3 months and 9 months after the intervention ends.
  Interventions: Behavioral: Next4You

INTERVENTIONS:
Behavioral: Next4You — Youth in the intervention arm will have access for four continuous weeks to a mobile intervention that covers topics related to communication, relationships, sexual wellness, contraception, respecting self and partners, and building wealth and wellness.

SUMMARY:
The purpose of the study is to rigorously evaluate Next4You, an innovative, fully mobile program featuring 6 content modules, each containing 8-10 microlessons intended to reduce rates of unintended pregnancy and sexually transmitted infections (STI) and increase essential knowledge, attitudes, and skills among young people aged 16-19 currently in the foster care system in California.

DETAILED DESCRIPTION:
Next4You will be tested using a randomized controlled trial (RCT) involving approximately 500-600 young people ages 16-19 with former or current experience in the California foster care system. Participants will complete an online screener that will assess eligibility (age, foster youth status, county of residence, English proficiency, and access to a device that is Wi-Fi or cellular enabled). Participants will be randomly assigned to receive access to the Next4You mobile platform and its microlessons and resources or a control website containing various health promotion materials. Participants in both conditions will have four consecutive weeks to explore the content on the platform (defined as the implementation period). Self-reported survey data related to attitudes, knowledge, and behavior around romantic relationships and sexual behavior are collected at baseline, as well as 3 months and 9 months after the intervention ends.

ELIGIBILITY:
Inclusion Criteria: Age, foster youth status, county of residence, English proficiency, access to a digital device that is Wi-Fi and/or cellular enabled -

Exclusion Criteria:

-

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-09-29 (Estimated)

PRIMARY OUTCOMES:
Prevalence of choosing abstinence or the use of other contraception and/or condoms if having vaginal or anal sex in the past 3 months | 3 months post-intervention
  Measured with single-item dichotomous measure of behavior analyzed individually to assess: any consensual vaginal sex in the past 3 months (main and casual sex partners); any consensual vaginal sex with a condom in the past 3 months (main and casual sex partners); any consensual vaginal sex with birth control other than condoms in the past 3 months (main and casual sex partners); consensual anal sex in the past 3 months (main and casual sex partners); and consensual anal sex with a condom in past 3 months (main and casual sex partners).

SECONDARY OUTCOMES:
Prevalence of choosing abstinence or the use of other contraception and/or condoms if having vaginal or anal sex in the past 3 months | 9 months post-intervention
  Measured with single-item dichotomous measure of behavior analyzed individually to assess: any consensual vaginal sex in the past 3 months (main and casual sex partners); any consensual vaginal sex with a condom in the past 3 months (main and casual sex partners); any consensual vaginal sex with birth control other than condoms in the past 3 months (main and casual sex partners); consensual anal sex in the past 3 months (main and casual sex partners); and consensual anal sex with a condom in past 3 months (main and casual sex partners).
Rates of condomless vaginal or anal sex | 3 months post-intervention
  Single measure constructed from number of times having consensual vaginal/anal sex in past 3 months; number of times using a condom during consensual vaginal/anal sex in past 3 months; number of times using birth control during consensual vaginal sex in past 3 months
Rates of condomless vaginal or anal sex | 9 months post-intervention
  Single measure constructed from number of times having consensual vaginal/anal sex in past 3 months; number of times using a condom during consensual vaginal/anal sex in past 3 months; number of times using birth control during consensual vaginal sex in past 3 months
Sexual consent self-efficacy | 3 months post-intervention
  A measure comprised of 35 questions from the Sexual Consent Scale (Humphreys & Brousseau, 2010) that measures perceived self-efficacy related to sexual consent at 3 months after intervention completion.
Sexual consent self-efficacy | 9 months post-intervention
  A measure comprised of 35 questions from the Sexual Consent Scale (Humphreys & Brousseau, 2010) that measures perceived self-efficacy related to sexual consent at 3 months after intervention completion.
Sexual communication self-efficacy | 3 months post-intervention
  A measure comprised of 20 questions from the Sexual Communication Self-Efficacy Scale (Quinn-Nilas et al., 2016) that measures perceived self-efficacy related to sexual communication at 3 months after intervention completion.
Sexual communication self-efficacy | 9 months post-intervention
  A measure comprised of 20 questions from the Sexual Communication Self-Efficacy Scale (Quinn-Nilas et al., 2016) that measures perceived self-efficacy related to sexual communication at 3 months after intervention completion.
Condom use attitudes/beliefs | 3 months post-intervention
  A measure comprised of 10 questions from the Multidimensional Condom Attitudes Scale (Helweg-Larsen & Collins, 1994) that measures attitudes related to condom use at 3 months after intervention completion.
Condom use attitudes/beliefs | 9 months post-intervention
  A measure comprised of 10 questions from the Multidimensional Condom Attitudes Scale (Helweg-Larsen & Collins, 1994) that measures attitudes related to condom use at 3 months after intervention completion.
Contraceptive use attitudes/beliefs | 3 months post-intervention
  A measure comprised of 11 measures from the Contraceptive Attitude Scale (Kyes, 1998) that measure attitudes related to contraceptive use at 3 months after intervention completion.
Contraceptive use attitudes/beliefs | 9 months post-intervention
  A measure comprised of 11 measures from the Contraceptive Attitude Scale (Kyes, 1998) that measure attitudes related to contraceptive use at 3 months after intervention completion.
Experiences with equity and power balance in relationships | 3 months post-intervention
  A measure comprised of the Relationship Control Subscale (15 questions) from the Sexual Relationship Power Scale (Pulerwitz et al., 2000) that measures equity and power balance in relationships at 3 months after intervention completion.
Experiences with equity and power balance in relationships | 9 months post-intervention
  A measure comprised of the Relationship Control Subscale (15 questions) from the Sexual Relationship Power Scale (Pulerwitz et al., 2000) that measures equity and power balance in relationships at 3 months after intervention completion.
Knowledge of health care rights and location of services | 3 months post-intervention
  A measure of the % of correct answers comprised from survey questions on knowledge of health care rights (Anderson et al., 2021; Coyle et al., 2021; Office of Management and Budget, n.d.) at 3 months after intervention completion.
Knowledge of health care rights and location of services | 9 months post-intervention
  A measure of the % of correct answers comprised from survey questions on knowledge of health care rights (Anderson et al., 2021; Coyle et al., 2021; Office of Management and Budget, n.d.) at 3 months after intervention completion.
Experience with condom use | 3 months post-intervention
  A count of condom issues experienced (derived from 8 condom experiences survey questions [Coyle et al., 2021]) at 3 months after intervention completion
Experience with condom use | 9 months post-intervention
  A count of condom issues experienced (derived from 8 condom experiences survey questions [Coyle et al., 2021]) at 3 months after intervention completion
Knowledge of educational rights and programs | 3 months post-intervention
  A measure of the % of correct answers comprised from 3 survey questions on awareness of rights and programs for youth in foster care going to college or trade school at 3 months after intervention completion
Knowledge of educational rights and programs | 9 months post-intervention
  A measure of the % of correct answers comprised from 3 survey questions on awareness of rights and programs for youth in foster care going to college or trade school at 3 months after intervention completion
Financial literacy knowledge | 3 months post-intervention
  A measure of the % of correct answers comprised from 3 survey questions on financial literacy knowledge at 3 months after intervention completion
Financial literacy knowledge | 9 months post-intervention
  A measure of the % of correct answers comprised from 3 survey questions on financial literacy knowledge at 3 months after intervention completion

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Anderson, PhD, Principal Investigator — ETR; Karin Coyle, PhD, Principal Investigator — ETR
Locations (1):
- RTI, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: No